CLINICAL TRIAL: NCT06518642
Title: Transcranial Direct Current Stimulation (tDCS) in Young Individuals with Major Depressive Disorder: a Literature Review and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCS_depression
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder (MDD); Youth; Transcranial Direct Current Stimulation (tDCS); Augmentative treatment; Young adults; Adolescent
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At the beginning of the stimulations sessions, participants receiving both the active and sham stimulation would experience a ramp-up in current from 0 to 2 mA, then the current would ramp down to 0 mA for participants receiving sham stimulation.
  Participants were told that they may experience sensations such as tingling, headache, or mild burning during the first 30 - 60 seconds of the stimulation session but that they may subside afterwards as they got used to it. In other words, participants would not be able to tell if diminishing of side effects were due to habituation (active tDCS) or ramping down of current (sham tDCS).
  Moreover, the stimulation mode of the tDCS device was pre-set by a the principal investigator, who was not involved in the stimulation delivery or outcome measurements, both of which were conducted by a research assistant who was blinded to the stimulation mode.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active stimulation (Experimental): A current strength of two mA will be consistently applied for 30 minutes, with 30 seconds of ramping up and ramping down periods.
  Interventions: Device: Sooma tDCS portable device - active stimulation
- sham stimulation (Sham Comparator): Current application will remain identical to the active stimulation, except that stimulation will be tampered off after 30 seconds. This duration (30 secs) was selected based on previous studies indicating that mild discomfort during active current application, such as tingling, would commonly be experienced up to 30 seconds only before subsiding
  Interventions: Device: Sooma tDCS portable device - sham stimulation

INTERVENTIONS:
Device: Sooma tDCS portable device - active stimulation — Treatment followed common tDCS protocol upon considering safety and tolerability, comprising five consecutive sessions in five days of 30-minute 2 mA tDCS. We utilized the Soterix Medical tDCS device (Soterix Medical, New York, NY, USA, Model 1x1 tDCS-CT) in the research lab and the Sooma Oy device (Sooma Depression Therapy Comfort, Helsinki, Finland) for patient self-administration.Sooma provided two of their portable tDCS devices for a brief period, including one customized sham device.Due to the limited availability of the Sooma devices, participants were randomly allocated to either the Sooma or. Due to the limited availability of the Sooma devices, participants were randomly allocated to either the Sooma or the Soterix device based on availability during their initial session. A current of 2 mA was applied with the anode positioned left DLPFC, corresponding to area F3 in the international 10-20 system. The cathode (reference electrode) was applied at the right dPLFC, F4.
  Arms: active stimulation
Device: Sooma tDCS portable device - sham stimulation — Sooma provided two of their portable tDCS devices for a brief period, including one customized sham device for effective blinding, distinguishable only by serial number and managed by an external data manager following the randomization sequence.To ensure blinding to the participant and their caregiver, at the beginning of the stimulation sessions, participants receiving both the active and sham stimulation would experience a ramp-up in current from 0 to 2 mA, and then the current would ramp down to 0 mA for participants receiving sham stimulation. Participants were told that they may experience sensations such as tingling, headache, or mild burning during the first 30-60 seconds of the stimulation session but that they may subside afterwards as they got used to it. In other words, participants would not be able to tell if diminishing of side effects were due to habituation (active tDCS) or ramping down of current (sham tDCS).
  Arms: sham stimulation

SUMMARY:
Objectives: (1) To assess the therapeutic effects of tDCS on improving depressive symptoms in young individuals with Major Depressive Disorder (MDD), relative to sham stimulation ; and (2) to evaluate the tolerability, and feasibility of tDCS in young individuals with Major Depressive Disorder, to explore the feasibility for a scale-up study.

Hypothesis: 1) we hypothesize the tDCS stimulation of the dorsolateral prefrontal cortex (dLPFC) will reduce symptoms of depression more than sham stimulation, demonstrated by significant difference in change of Hamilton Depression Rating Scale (HDRS) and 2) tDCS active stimulation of the dLPFC will be tolerable and feasible among patients with MDD, as demonstrated by minimal adverse effects measured in the Adverse Events Questionnaire, adherence (with reasons of drop out), their motivation and enjoyment to participate in the study .

DETAILED DESCRIPTION:
The incidence of probable depression during the fifth peak of COVID-19 was 24.6%, within the HK population, with the youths having experienced a disproportionately higher rate. A recent epidemiology survey conducted in HK revealed the 12-month prevalence of suicidal ideation among young individuals above secondary school age to be an alarming 8.4%. While guidelines and RCTs support the use of medication and psychotherapy as a standalone or combination treatments for major depressive disorder (MDD) in youths, a large proportion do not respond to either medication or psychotherapy. There is therefore an unmet need for new, effective treatment options for depression that can be tolerated by young individuals. Transcranial direct current simulation (tDCS) has its acute-effect is physiological change that reduces the threshold of membrane polarisation and increased the synaptic excitability. A handful of studies suggested that anodal stimulation of the dorsal lateral prefrontal cortex (DLPFC) is effective in reducing depressive symptoms in adults, however, whether similar effects applies to youth remains unknown. tDCS is portable, relatively inexpensive, and easy to use, proving to be very safe and tolerable for young individuals with minimal and temporary side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with major depressive disorder (MDD) according to the Structured Clinical Interview for DSM-5, Clinical Version (SCID-DSM-5, CV)
* Scored ≥ 14 (i.e., at least mild to moderate depression on the 17-item Hamilton Depression Rating Scale (HDRS) at screening and at baseline;
* Right handedness;
* Stable dosage of antidepressants or other treatments for depression in recent 4 weeks; and
* Can read and write Chinese.

Exclusion Criteria:

* History of significant head trauma, neurological disorders (e.g., epilepsy), seizures;
* First degree relative with epilepsy;
* Concomitant unstable medical conditions; major neurological conditions;
* Comorbid disorders listed in the DSM-V, e.g., schizophrenia, substance use disorder, mental retardation, etc.;
* Pregnancy, lactating women, or women planning pregnancy;
* Device or metal clips on or inside the skull, cardiac pacemaker;
* Inability to provide informed consent.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) - 17 items | T0 (baseline); T1 (immedately after intervention)
  Measuring depressive symptoms, score ranges from 0 (minimum) to 53 (maximum); higher score indicates more severe depressive symptoms.

SECONDARY OUTCOMES:
Social and Occupational Functioning Assessment scale (SOFAS) | T0 (baseline); T1 (immedately after intervention)
  Measures social and occupational functioning across work functioning, independent functioning, immediate and extended social network functioning; score ranges from 0 (minimum) to 100 (maximum), higher score indicates higher social and occupational functioning ability.
Role Functioning Scale (RFS) | T0 (baseline); T1 (immedately after intervention)
  Measures role functioning in four areas: work productivity, independent living, immediate and extended social network relationships; score ranges from 0 (minimum) to 7 (maximum) on each aspect, higher score indicates better role functioning
Global Functioning: Social Scale and Role Scale | T0 (baseline); T1 (immedately after intervention)
  Measures social and role functioning; score ranges from 1 (minimum) to 10 (maximum); higher score indicates better social/role functioning
Short Form Health Survey (SF-12) | T0 (baseline); T1 (immedately after intervention)
  Short-form measure of health status with 12 questions.
Clinical Global Impression Scale | T1 (immedately after intervention)
  Measures the severity of illness and global improvement following an intervention; scores ranges from 1 (normal/very much improved) to 7 (most severely ill/very much worse), with higher scores indicating worse outcome.
Beck Scale of Suicidal Ideation. | T0 (baseline); T1 (immedately after intervention)
  Measures self-reported suicidal ideation; score ranges from 0 (minimum) to 38 (maximum), with higher scores indicating a greater risk of suicide.
Visual Analog Scale (VAS) | T0 (baseline); T1 (immedately after intervention)
  Two VASs were used to measure motivation and willingness during intervention. Each VAS contains a scale of 0 (minimum) to 10 (maximum) with higher scores indicating more
Chinese version of the Snaith-Hamilton Pleasure Scale (C-SHAPS) | T0 (baseline); T1 (immedately after intervention)
  Gold standard, self-rated scale measuring anhedonia symptoms. Each item ranges from 0 to 3, hence total score ranges from 0 (minimum) to 42 (maximum) with higher scores indicating more anhedonic symptoms
Chinese version of the Dimensional Anhedonia Rating Scale (C-DARS) | T0 (baseline); T1 (immedately after intervention)
  17-item self-rated questionnaire measuring anhedonia symptoms. Each item ranges from 0 to 4, hence total score ranges from 0 (minimum) to 68 (maximum) with higher scores indicating lower levels of anhedonia symptoms
Adherence rate to the participation of the tDCS study | from T0 (baseline) to T1 (immedately after intervention)
  Adherence rate of full participation in each tDCS session; and the reason of skipping the tDCS session if any

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong